CLINICAL TRIAL: NCT06564935
Title: Preoperative Oral Heptaminol Hydrochloride in Preventing Hypotension After Spinal Anesthesia in Lower Limb Surgeries With Tourniquet: A Randomized Controlled Trial
Brief Title: Preoperative Oral Heptaminol Hydrochloride in Preventing Hypotension After Spinal Anesthesia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdElKhalik Mahmoud Shaban, Lecturer of anaesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MS-186-2024
Record Dates: First submitted 2024-08-16; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Hypotension After Spinal Anesthesia
MeSH Terms: interventions — Heptaminol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heptaminol hydrochloride group (Active Comparator)
  Interventions: Drug: Heptaminol Hydrochloride
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Heptaminol Hydrochloride — heptaminol hydrochloride will be administrated in its solution form 4ml/kg. The mean dose used will be 25 drops = 150 mg and will be given 1.5 to 2 hours before spinal anesthesia
  Arms: Heptaminol hydrochloride group
Drug: Placebo — Placebo drops (identical to heptaminol drops, prepared by the hospital pharmacy) will be administered 1.5 to 2 hours before spinal anesthesia.
  Arms: Placebo group

SUMMARY:
Methodologies and approaches have been implemented with differing degrees of success to prevent neuraxial hypotension. Currently utilized approaches to prevent hypotension during spinal anesthetic administration consist of physical precautions such as leg restraints and compression hosiery, as well as sympathomimetic medications Through a competitive inhibition of noradrenaline uptake, heptaminol hydrochloride prevented orthostatic hypotension and increased the plasma concentration of noradrenaline. This inhibitory effect might account for a portion of the antihypotensive effect After thorough research of the literature, studies evaluating the role of preoperative oral heptaminol hydrochloride in preventing hypotension after spinal anesthesia in lower limb surgeries with tourniquets are lacking.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 50 years old.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I-II.
* Undergoing elective orthopedic lower limb operations with a tourniquet or plastic surgeries under spinal anesthesia.

Exclusion Criteria:

* Patient refusal.
* History of hypertension, cardiovascular [disorders of the heart and blood vessels and including coronary heart disease, rheumatic heart disease and other conditions], and cerebrovascular diseases [conditions that affect blood flow and the blood vessels in the brain. Problems with blood flow may occur from blood vessel narrowing (stenosis), clot formation (thrombosis), artery blockage (embolism), or blood vessel rupture (hemorrhage)].
* Baseline SBP >160 mm Hg before administration of the drug.
* Any contraindications to spinal anesthesia such as coagulopathy, local skin infection, swelling, trauma, or deformity.
* Medical conditions, which release vasoconstrictors such as pheochromocytoma.
* Patients taking vasoconstrictors or uncorrected tachyarrhythmia.
* History of drug allergy.
* Psychiatric, neuromuscular disorder, major systemic diseases.
* Pregnancy or lactating women.
* Inadequate effect of spinal anesthesia or supplemented with other types of anesthesia.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Hypotension | It will be assessed in the first 20 minutes after spinal anaesthesia
  The occurrence of hypotension is defined as SBP <90 mm Hg or <80% of baseline, after spinal anesthesia. Our hypotension outcome was a binary event (yes/no) defined as the occurrence of at least 1 episode for a patient below either threshold, versus none, across the repeated measurements.

SECONDARY OUTCOMES:
Changes in mean arterial blood pressure after spinal anesthesia | Every 5 minutes in the first 20 minutes after spinal anesthesia then every 15 minutes until the end of operation assessed up to 3 hours after spinal anesthesia
  Duration measurement of serial changes in mean arterial blood pressure after spinal anesthesia
Changes in heart rate after spinal anesthesia | Every 5 minutes in the first 20 minutes after spinal anesthesia then every 15 minutes until the end of operation assessed up to 3 hours after spinal anesthesia
  Duration measurement of serial changes in heart rate after spinal anesthesia

OTHER OUTCOMES:
Requirements of ephedrine | From the time of intrathecal injection of the anesthetic drug until the end of operation after spinal anesthesia assessed up to 3 hours after spinal anesthesia
  The total requirements of ephedrine to treat hypotension
Requirements of Atropine | From the time of intrathecal injection of the anesthetic drug until the end of operation after spinal anesthesia assessed up to 3 hours after spinal anesthesia
  The total requirements of ephedrine to treat bradycardia